CLINICAL TRIAL: NCT05064241
Title: Investigations of Barriers and Methods to Overcome Barriers to Access Genetic Medicine
Brief Title: Overcoming Barriers to Accessing Genetic Medicine
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Principal Investigator, Catherine Brownstein, Assistant Professor, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: P00039779
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Genetic Disease; Genetic Predisposition
MeSH Terms: conditions — Genetic Diseases, Inborn; Genetic Predisposition to Disease

STUDY DESIGN:
Intervention Model Description: One group has access to a genetic counselor answering their questions, another group has peer-to-peer conversation. However, at the end of the study, the genetic counselor will answer the questions asked in the peer-to-peer discussion board.
Who Masked: Participant
Masking Description: Participants will not be told which discussion board they are randomized to. However, they may possibly discover that one board has a genetic counselor, and the other does not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Advisory Board (Experimental): Participants have access to a genetic counselor to answer their questions on accessing genetic medicine.
  Interventions: Other: Access to Genetic Counselor for answering questions
- Virtual Peer-to-Peer Discussion Board (No Intervention): Participants answer each others' questions on the topic of accessing genetic medicine.

INTERVENTIONS:
Other: Access to Genetic Counselor for answering questions — A genetic counselor answers questions posed by participants in the intervention arm on how to access genetic medicine. At the end of the study, the number of participants who were able to access genetic medicine will be assessed
  Arms: Virtual Advisory Board

SUMMARY:
To learn about patient barriers to accessing genetic medicine, we will analyze anonymous posts from a membership-based online community [Inspire.com], and investigate how these barriers differ for various populations. We will then test whether these barriers can be addressed by providing online access to a genetic counselor to answer patient questions for one group of patients (virtual advisory board group) and compare to that of a control group who does not have access to a genetic counselor (virtual peer-to-peer board group).

DETAILED DESCRIPTION:
Genomic medicine has the potential to advance diagnoses, predict risk, support prevention efforts, and inform treatment decision-making. Though technologies for measuring genetic variants have improved and become more cost-effective, clinical integration of genomic medicine has been surprisingly slow. For genomic medicine to be successfully implemented across specialties and across demographics, the systemic barriers that patients experience need to be identified and addressed.

Online health support is becoming an increasingly important part of healthcare as more patients use digital health networks. In the first part of this study, an analysis of online communication in a membership-based online support community [Inspire.com] will identify systemic, structural and individual barriers to accessing genomic medicine. A genetic counselor will be informed to these results and will be part of the intervention arm of the study.

To assess the extent to which online health networks can directly help genomic medicine implementation, participants will join one of two Virtual Discussion Boards (a Virtual Advisory Board and a Virtual Peer-to-Peer Discussion Board). In the intervention arm, the Virtual Advisory Board will have a genetic counselor answer patient questions online about genomic medicine once every week for a period of three months. In the control arm, participants will answer and comment on each others' questions in the Virtual Peer-to-Peer Discussion Board. We hypothesize that after six months, patients who participate in the Virtual Advisory Board are more likely to self-report receiving genomic medicine than those in the control arm. After completion of the study, participants in the Peer-to-Peer Discussion Board, we will give online access to the genetic counselor to answer any questions

ELIGIBILITY:
Inclusion Criteria:

Member of Inspire.com Genetic disease Genetic predisposition to disease -

Exclusion Criteria:

Not member of Inspire.com No genetic disease No genetic predisposition to disease

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Qualitative self-report of referrals for clinical genetic services | 6 months
  Percentage of participants with self-report of referrals for clinical genetic services

SECONDARY OUTCOMES:
Qualitative self-report of specific barriers to the participant accessing genomic medicine | 6 months
  The ability for a participant to articulate the barriers to them accessing genetic medicine
Self-report of specific behaviors to overcome barriers to accessing genetic medicine | 6 months
  Qualitative assessment of ability for a participant to self-report performing behaviors to overcome barriers to accessing genetic medicine.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
We will share aggregated and de-identified data as requested in accordance with our IRB protocol.